CLINICAL TRIAL: NCT02771951
Title: Clinical/Behavioral Approach to Overweight in Latino Youth: Luces de Cambio
Brief Title: Clinical/Behavioral Approach to Overweight in Latino Youth
Acronym: Luces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, John Elder, Distinguished Professor of Public Health; and Adjunct Professor of Family and Precentive Medicine, UCSD, San Diego State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: SanDiegoStateU
Record Dates: First submitted 2016-05-09; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Overweight; Pediatric Obesity
Keywords: Childhood; Obesity
MeSH Terms: conditions — Overweight; Pediatric Obesity; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Special Intervention (Experimental): Study participants randomized to receive Special Intervention receive a series of 7 group classes taught by trained clinic health educators; a series of phone calls; clinical visits with a mid-level provider; and a series of 6 booster group classes over 1 year.
  Interventions: Behavioral: "Lights of Change"
- Usual Care (Placebo Comparator): Study participants randomized to receive Usual Care receive up to 2 visits with a usual care health educator over 1 year.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: "Lights of Change"
  Arms: Special Intervention
Behavioral: Usual Care
  Arms: Usual Care

SUMMARY:
This randomized controlled trial tests the efficacy of a culturally and linguistically appropriate, evidence-based intervention to slow weight gain or promote weight loss among overweight 6-9 year old Mexican-American children.

DETAILED DESCRIPTION:
Overweight and obesity is a serious problem for Mexican-American children, due in part to poverty, acculturation, genetic predisposition or other factors. Clinic-based weight control studies have shown promise, but often include convenience samples with few or no Latino children. This randomized controlled trial tests the efficacy of a culturally and linguistically appropriate, evidence-based intervention to lower Body Mass Index (BMI) or slow weight gain among overweight 6-9 year old Mexican-American children randomly sampled from a large (36,192 pediatric patients) community clinic providing services to low and medium income families in a US-Mexico border community (San Ysidro, CA). Intervention and measurement design and selection are based on a "Socioecological Model for Latino Health Promotion". Children and their parents will be randomly assigned to either a Special Intervention (SI) or Usual Care (UC) group. The SI group will participate in the following behavior change activities based on Prevention Plus and Structured Weight Management approaches:

1. classes providing culturally-sensitive health education regarding healthy eating, increasing physical activity, decreasing sedentary behaviors, and effective parenting behaviors to model and reinforce children's health behaviors, instruction on how to modify both social and structural aspects of the home environment, and skills-building to navigate community resources;
2. clinical visits with a Health Educator and Mid-Level Provider (MLP);
3. family visits with primary care providers (PCP); and
4. phone calls to reinforce goal setting.

The UC group will receive standard health education for childhood obesity already provided by the community clinic. The primary outcome for the study is child BMI, which along with other changes in physical outcomes, child health behaviors and parenting behaviors will be evaluated at four time-points (baseline, 6-, 12-, and 18-months). The primary hypothesis is that the SI group will demonstrate lower mean BMI than the UC group at the end of a 6 month intervention with a maximum difference occurring at 12 months, and will sustain this difference for an additional six months (18 months after baseline). Secondary aims include examining intervention effects on children's energy balance, physical activity levels, sedentary behavior and parenting strategies related to their children's health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Latino
* Have made a clinic visit within past 24 months prior to enrollment in study
* Have a BMI % for age/gender between 75 - 99.9th
* Plan on living in target area for following 18 months
* Have transportation to participating clinic

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 297 (Actual)
Dates: Start 2010-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Behavioral and Community Health at San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No